CLINICAL TRIAL: NCT06447038
Title: Pilot Study for the Early Detection of Chronic Kidney Disease, Non-Dialysis Objective (NDO).
Acronym: NDO
Status: Enrolling by invitation | Type: Observational
Sponsor: Hospital Universitario de Burgos (Other)
Responsible Party: Principal Investigator, Didier Sánchez OSpina, Doctor investigator, Hospital Universitario de Burgos
Other Study IDs: OND 01
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Chronic Kidney Disease (CKD)
Keywords: Epidemiology.; Chronic kidney disease.; Primary care.; Cardiovascular risk factors.
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Population: Population of the city of Burgos > 18 years old.
  Interventions: Diagnostic Test: albumin creatinine ratio

INTERVENTIONS:
Diagnostic Test: albumin creatinine ratio — Albumin creatinine ratio, this test is routinely performed in urine.

SUMMARY:
Chronic kidney disease (CKD) is a significant public health problem worldwide, affecting more than 10% of the Spanish population. Early detection is considered a top healthcare priority to establish strategies for preventing progression to more advanced stages of the disease and its complications. Additionally, CKD is associated with high comorbidity, poor prognosis, and substantial resource consumption within the healthcare system. In this context, albuminuria may be a more sensitive marker of CKD than reduced glomerular filtration rate (GFR), and it is also considered an indicator of not only renal damage but also "systemic damage" (generalized endothelial dysfunction, arterial remodeling, and increased cardiovascular risk) beyond the kidney. Furthermore, the reduction of proteinuria/albuminuria is clearly associated with a slower progression of CKD, making its reduction a therapeutic goal as well. Given this importance, this protocol aims to determine the urine albumin/creatinine ratio in all patients over 18 years old who visit their primary care physician in the province of Burgos, Spain, and require a blood test related to their reason for consultation.

DETAILED DESCRIPTION:
This is a protocol in which we seek to identify those patients with alterations incipient renal failure by determining the albumin/creatinine ratio in urine, test that is currently performed routinely in different groups of patients. By For this reason, the implementation of the non-dialysis objective protocol hopes to be implemented standardized form in patients who go to their primary attention doctor in the province of Burgos to later be extended to the entire Castilla y Leon community.

.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18 years

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of the city of Burgos, Spain who go to their primary doctor.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Albumin creatinine ratio. | 01/02/2024 al 01/12/2024
  Determination of albuminuria in urine.

CONTACTS AND LOCATIONS:
Overall Officials: Maria J Izquierdo Ortiz, Doctor, Study Director — HUBU; Emilio J Gonzalez Parra, Doctor, Principal Investigator — HUBU; Sebastian Mas Fontao, Doctor, Principal Investigator — HUBU; Maria Martin Palencia, Doctor, Principal Investigator — HUBU; Didier Sanchez, Doctor, Study Director — HUBU
Locations (1):
- Maria J Izquierdo, Burgos, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750